CLINICAL TRIAL: NCT02174393
Title: Efficacy of Combination Therapy With Microneedling and the Universal Peel For Acne Scarring in Skin Types III-VI
Brief Title: Microneedling Plus the Universal Peel For Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Collaborators: Topix Pharmaceuticals (Unknown); Eclipse Aesthetics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-14-555
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Acne Scarring
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microneedling Plus Universal Peel (Experimental): (1) Microneedling treatment by the MicroPen with a Post-Microneedling Skin Care Regimen and the (2) Universal Peel by Topix with a Post-Universal Peel Skin Care Regimen will both be performed on a monthly basis for a total of three treatment sessions each.
  Microneedling will be done on Study Weeks 1, 5, and 9. Universal Peel will be done on Study Weeks 3, 7, and 11.
  Interventions: Drug: Universal Peel; Procedure: Microneedling; Drug: Post-Microneedling Skin Care; Drug: Post-Universal Peel Skin Care

INTERVENTIONS:
Drug: Universal Peel — Universal Peel: is a chemical peel consisting of a mild acid solution. (5 min Peel and 5 min Retinol)
Procedure: Microneedling — Microneedling: is a device for all skin types that creates micro "injuries" in the dermis (layer of the skin underneath the outermost layer) in an attempt to trigger new collagen (natural component of skin tissue) production for smoother, firmer and younger-looking skin.
  For this protocol, the needle depth will be increased over the 3 sessions:
  Forehead: 0.75 mm, 0.85 mm, 1.0 mm. Cheeks/Chin: 1.0 mm, 1.5 mm, 2.0 mm.
  Each Session: Microneedling procedure on Day 1, followed by skin care regimen
Drug: Post-Microneedling Skin Care — On Day 1 (after Microneedling procedure):
  * Gentle Antioxidant Soothing Cleanser daily
  * Soothing Recovery Ointment and Sheer Physical Sunscreen
  On Day 2-7:
  * AM: Physical sheer sunscreen and recovery ointment
  * PM: Retinol/Vitamin C in the evening and soothing recovery ointment
  On Day 7:
  * AM: BD Hydrating Day/Night Cream
  * PM: Retinol and Vitamin C and the BD Hydrating Day/Night Cream (if necessary)
Drug: Post-Universal Peel Skin Care — * Gentle Antioxidant Soothing Cleanser daily
  * Physical Sunscreen daily
  * Soothing recovery ointment fortified with silver only when peeling occurs
  * After completely peeling, vitamin c product in the morning and the retinol in the evening

SUMMARY:
Acne is a prevalent disorder mostly witnessed in adolescents, but can be seen in adults. Early treatment is imperative to reduce acne scarring which can appear with atrophic lesions, and depending on the skin type, significant erythema (redness) or post-inflammatory hyperpigmentation. A multi-modality approach to treatment is necessary when dealing with the aforementioned types of lesions. Pharmacologic management is essential, but safe procedural therapies are also necessary specifically with darker skinned individuals.

Percutaneous collagen induction therapy (PCIT) is a non-invasive treatment achieved by using a micro-needling device, which is safe and effective in causing "micro-wounds" into the dermis thereby initiating wound healing followed by collagen production. This is an ideal treatment for acne scarring, re-texturizing of the skin, and hyperpigmentation for all skin types . Currently there are very few studies evaluating the safety and efficacy of microneedling and chemical peels in skin types III-VI.

The aim of this study is to evaluate the effects of the combination of microneedling and chemical peel for the treatment of acne scars in skin types III-VI.

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 and < 60 years of age.
* Subject has skin type III, IV, V, or VI as defined by the Fitzpatrick Classification Scale.
* Subject has acne scarring as defined by the Goodman and Baron Grading System.

Exclusion Criteria:

* Subject currently has moderate to severe acne on the face.
* Subject has an active infection.
* Subject is pregnant or lactating.
* Subject has a history of a bleeding disorder.
* Subject is taking an anti-coagulant.
* Subject has a history of keloidal tendency.
* Subject has received ablative or non-ablative laser treatments in the previous 6 months.
* Subject has taken Accutane within the previous 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement in the appearance of acne scarring as measured by The Goodman and Baron Grading Scale. | 6 months
  The scale will be completed at every office visit over the 6 month study (Baseline, Weeks 1, 3, 5, 7, 9, 11, and 17).
Improvement in the appearance of acne scarring as measured by the 4 Point Scar Scale. | 6 Months
  The scale will be completed at each office visit during the 6 month study (Baseline, Weeks 1, 3, 5, 7, 9, 11, and 17).
Improvement in the appearance of acne scarring as measured by the Global Assessment. | 6 months
  The Global Assessment of Improvement will be completed at Week 17.

SECONDARY OUTCOMES:
Improvement in the appearance of acne scarring as subjectively measured through digital pictures. | 6 months
  Pictures of the subject will be taken by the Principal Investigator at every office visit during the 6 month study (Baseline, Weeks 1, 3, 5, 7, 9, 11, and 17).
Patient-reported improvement in the appearance of acne scarring as measured by the Cardiff Index. | 6 months
  The Cardiff Index will be completed at Baseline and Week 17.
Patient reported improvement in appearance of acne scarring a measured by pre and post-treatment questionnaires. | 6 months
  Subject will complete a pre-treatment questionnaire at Baseline and post-treatment questionnaires at Weeks 7 and 17.

CONTACTS AND LOCATIONS:
Overall Officials: Naana Boakye, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Bergen Dermatology, Englewood Cliffs, New Jersey, United States